CLINICAL TRIAL: NCT03690752
Title: Adherence to Walking on an Alter G Anti-Gravity Treadmill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2017-275
Record Dates: First submitted 2018-09-25; First posted 2018-10-01 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Severe Obesity
Keywords: Obesity; Alter-G Anti-Gravity Treadmill; 6-minute walk test; timed up and go test; physical activity enjoyment; pain
MeSH Terms: conditions — Obesity, Morbid; Obesity; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- weighted (Sham Comparator): The weighted group uses the same Alter-G Treadmill as the unweighted group but were not allowed to use the unweighting function of the treadmill.
  Intervention: unweighting using Alter-G Anti-Gravity Treadmill
  Interventions: Device: normal weight using Alter-G Anti-Gravity Treadmill
- unweighted (Experimental): The unweighted group uses the same Alter-G Anti-Gravity Treadmill as the weight group but is allowed to adjust their weight using the weight control feature.
  Intervention: normal weight using Alter-G Anti-Gravity Treadmill
  Interventions: Device: unweighting using Alter-G Anti-Gravity Treadmill

INTERVENTIONS:
Device: unweighting using Alter-G Anti-Gravity Treadmill — The unweighted group (experimental) is allowed to self-select a comfortable unweighting using the weight control feature on the Alter-G Anti-Gravity Treadmill. Both groups use the same Alter-G Anti-Gravity Treadmill and both groups are about to self-select speed, incline, and duration.
  Other Names: Lower body positive pressure
  Arms: unweighted
Device: normal weight using Alter-G Anti-Gravity Treadmill — The weighted (control) group will walk at 100% their body weight using the Alter-G Anti-Gravity Treadmill. Both groups use the same Alter-G Anti-Gravity Treadmill and both groups are about to self-select speed, incline, and duration.
  Other Names: lower body positive pressure
  Arms: weighted

SUMMARY:
Several barriers to exercise are present that need to be addressed. Morbidly obese individuals experience more skin friction, urinary stress incontinence, knee pain, low back pain, and hip arthritis than the lean population, which may significantly impair their ability to adhere to an exercise regimen (6). Obesity and overweight also contribute to greater perceived effort, oxygen uptake, and less pleasure during treadmill exercise sessions (7). Recent theories suggest that a negative experience associated with exercise can significantly reduce the likelihood of engaging in future exercise sessions (8). Therefore, tools to reduce these barriers may improve outcomes for exercise-based interventions for morbid obesity.

The Alter-G, an antigravity treadmill that alleviates body weight while subjects exercise, has potential to reduce pain and exertion during exercise. Overall, these treadmills have been found to be effective for weight loss in obese populations (10). However, although evidence suggests that the Alter-G would reduce pain and exertion, the effect of the Alter-G treadmill on exercise adherence in morbidly obese populations has not been studied.

The hypothesis is that the adherence to and progression of the exercise routine of participants walking at a reduced percentage of their body weight will increase relative to those who must exercise at 100% of their body weight.

A secondary hypothesis is that participants who use the Alter-G with the anti-gravity function will experience less pain and perceived exertion during exercise compared to those who exercise at 100% of their body weight.

Finally, the investigators hypothesize that increased exercise adherence in those using the anti-gravity function of the Alter-G will lead to increased fitness and improved muscle function.

DETAILED DESCRIPTION:
Screening

* A self-administered pre-participation health screening questionnaire (which contains physical activity readiness questionnaire (PAR-Q) questionnaire) will be used to ensure the eligibility for the study.
* Consent Form

III.) Exercise Protocol:

Scheduling:

Before beginning phases of the program, participants will be shown a physical calendar that will be located in the same room as the treadmill. They will be able to come in and select time slots in which they are available. Once a time slot has been filled it may not be reserved by another participant. If a schedule change is needed the participants will be allowed to come in and change it on the calendar and reserve an open time slot, while removing their name from the one they will be missing, or email the study coordinator and have a student or faculty member on the project change it for them.

Participants will take part in information and orientation session before scheduling begins. Informed consent will be obtained during this time, and this information session will serve as an overview of the program, and will introduce them to the Alter-G antigravity treadmill. They will be informed on how this exercise program will proceed, and will be told what to expect. Orientation Session During the orientation session, first measure blood pressure and resting heart rate as a final screening measure, and make sure it is not above 140/90 or heart rate (HR) of 90. The investigator will then review the study brochure with participants and complete informed consent. Once informed consent is obtained, participants will randomize them perform the sit-to-stand assessment followed by the 6 minute walk assessment then introduce them to the treadmill according to the following protocols:

Unweighting group:

1. Determine the participant's age-adjusted heart rate maximum.
2. Help the participant put on the polar strap heart rate monitor.
3. Help them select the shorts that fit them. Shorts should come up to the mid-hip, and should fit tightly around the thighs to make an air-tight seal.
4. Help the participant step into the treadmill.
5. Pull the bars up to mid-hip height, to be in line with the shorts. Lock the treadmill in place for the participant. Note down at which height the machine was at.
6. Help the participant zip the shorts in, and calibrate the treadmill.
7. Have the participant begin walking on the treadmill at a slow, comfortable pace. Let them get settled here and walk for 2 minutes.
8. Let them know the investigator will be bringing it down to 80% of their body weight, and do so. Let them remain at this % body weight for one minute.
9. Bring them down to 65% body weight. Allow them to adjust the pace of walking until they are comfortable, if needed, and remain there for one minute.
10. Bring them down to 50% body weight. Allow them to adjust the pace of walking until they are comfortable, if needed, and remain there for one minute.
11. Instruct the participant to select the unweighting that they feel comfortable and as pain-free as 10.1 possible, that still feels challenging. Help them adjust the pace of their walking as needed, as they find this ideal % body weight.
12. Let them walk at this unweighting at the pace they are comfortable for 5 minutes, and determine if their heart rate reaches 50-70% age-predicted maximum. If it does not, help them increase the pace until they do reach this heart rate range. If they still do not enter that range after another 3 minutes walking at the faster pace, ask the participant to either increase their pace again or increase their weight until they do. Note down the % body weight and pace, as this will be their baseline to work from throughout the program.

Control Group:

1. Determine the participant's age-adjusted heart rate maximum.
2. Help the participant put on the polar strap heart rate monitor.
3. Help them select the shorts that fit them. Shorts should come up to the mid-hip, and should fit tightly around the thighs to make an air-tight seal.
4. Help the participant step into the treadmill.
5. Pull the bars up to mid-hip height, to be in line with the shorts. Lock the treadmill in place for the participant. Note down at which height the machine was locked at.
6. Help the participant zip the shorts in, and calibrate the treadmill.
7. Have the participant begin walking on the treadmill at a slow, comfortable pace. Let them get settled here and walk for 2 minutes.
8. Work with the participant to find a pace that gets them to 50-70% of the age-adjusted heart rate maximum. This will be their baseline pace for the program. Before the participant leaves their orientation session, obtain their baseline body composition using the bioimpedance analysis (BIA) scale, an ultrasound of the thigh, their baseline health-related quality of life and history of join pain. Phase I [Weeks 1 - 2]

Goals:

* Begin program
* Explain and emphasize the individualized goals for each participant
* Record resting BP, HR, age-predicted max heart rate
* Start with a 5-10 minute warm up
* Monitor HR, rate of perceived excretion (RPE), and McGill Pain Inventory throughout exercise session

  o During the first session, as participants are walking on treadmill, the investigator will be recording these measurements.
* Allow participants to self-select an intensity that is comfortable for each subject individually while encouraging them to come in at least 3 days a week and work for at least 30 minutes a day.
* Should aim to reach a moderate intensity during the active part of the program (~50-70 % age-predicted max heart rate, 12-13 RPE on a Borg Scale, 2.0-4.0 mph).
* Reduce intensity for a 5-10 minute cool-down at the end

Treatment:

* The treatment group should walk at individualized percentage of body weight that was established during their orientation session for at least 30 minutes where there is reduced pain, or an absence of pain. Phase II [Weeks 2 - 16]

Goals:

* Continue program
* Start with a 5-10 minute warm up.
* Record HR, RPE, every session, and BP, and McGill Pain Inventory once per week.
* Meet with each participant individually every two weeks to:

  o Encourage participants to increase workload intensity and aim for longer and more frequent sessions on the treadmill.
* For those who met the 30 minutes for 3 days, they will be encouraged to increase their speed, duration, and/or incline.
* For those who were unable to meet the 30 min/3 day minimum they will be given advice on how to meet this minimum time. These meetings will serve as troubleshooting sessions.

  o Answer any questions the participants may have.
* Address any questions, comments, concerns, and complaints.
* Reduce intensity for a 5-10 minute cool-down at end of each session.

Final Session:

1. During the final exercise session, have the participant perform the sit-to-stand and 6 minute walk assessments then have the participant perform their baseline exercise session. Record their heart rate and RPE during this session to be compared to HR and RPE during the first session.
2. Ask the participant to fill out health-related quality of life questionnaire.
3. Measure participant's final body composition on the BIA scale and muscle thickness/ intramuscular fat content using ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* 20-55 years
* 30 and up BMI
* Passing PAR-Q

Exclusion Criteria:

* diagnosed metabolic, cardiovascular, or renal disease, or symptoms of these diseases
* participates in regular physical activity
* experienced a large fluctuation in body weight
* pregnant
* blood pressure more than 140/90
* resting heart rate more than 100 per minute
* hip size greater than 58" or less than 18.5"
* weight more than 400 lb
* height less than 4' 8"

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-09-09 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Adherence differences between groups | 12 weeks
  compare adherence to exercise during a 12 week program between the participants in the control and experimental groups using percentage of visit attended and minutes completed each week.

SECONDARY OUTCOMES:
difference in change in physical activity enjoyment between groups | From the first pre to post visits, assessed for 12 weeks
  difference in change for physical activity enjoyment is assessed using the physical activity enjoyment scale which is administered the first and last visits of the participants. The scale consist of 18 questions and the total will be obtained from the pre and post visits. The results from the post visit will have the first visit subtracted and the change will be the outcome.
difference in change in quality of life between groups | From pre to post visits, assessed for 12 weeks
  Quality of life is recorded using the WHOQOL-BREF questionnaire. The questionnaire consist of a total and four domains which include physical health, psychological, social relationships, and environmental. The questionnaire is administered pre and post and the change is post subtracted by pre.
difference in change in self-efficacy between groups | From pre to post visits, assessed for 12 weeks
  Self-efficacy is recorded using the self-efficacy questionnaire. The questionnaire consist of five questions and is administered pre and post with the change deriving from post minus pre.
difference in change in rate of perceived excursion between groups | From pre to post visits, assessed for 12 weeks
  Rate of perceived excursion (RPE) is collected during each exercise session. RPE will be averaged for each exercise session for each participant, then averaged over the 12 weeks and compared between groups.
difference in change in pain between groups | From pre to post visits, assessed for 12 weeks
  Pain is assessed using the Short Form McGill pain questionnaire.
difference in subjective pain between groups | From pre to post visits, assessed for 12 weeks
  Subjective pain is collected during each exercise session. Subjective pain will be averaged for each exercise session for each participant, then averaged over the 12 weeks and compared between groups.
difference in change in 6-minute walk test between groups | From pre to post visits, assessed for 12 weeks
  The 6-minute walk test is administered pre and post and change is done by subtracting the pre from the post.
difference in change in timed up and go test between groups | From pre to post visits, assessed for 12 weeks
  The timed up and go test is administered pre and post and change is done by subtracting the pre from the post.
difference in change in heart rate during the 6-minute walk test between groups | From pre to post visits, assessed for 12 weeks
  During the 6-minute walk test heart rate is measured at 2,4,and 6 minutes. Each individuals heart rates during the pre test will be averaged then those totals will be averaged for each group, same for the post test. The change will be post minus pre groups averages.
difference in change in blood pressure during the 6-minute walk test between groups | From pre to post visits, assessed for 12 weeks
  Blood pressure is administered right after completing the 6-minute walk test. The average blood pressure for each group for pre and post will be used to find change (post minus pre).
difference in change in rate of perceived excursion during the 6-minute walk test between groups | From pre to post visits, assessed for 12 weeks
  Rate of perceived excursion (RPE) is administered right after completing the 6-minute walk test. The average RPE is collected for each group for pre and post measurements, then post minus pre will get change in RPE.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Dhurandhar, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Department of Kinesiology and Sport Managment, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Once data collection is complete.
Supporting Information: Study Protocol, Analytic Code
Time Frame: After manuscript describing the study is released then the study protocol and analytic code will be shared.
Access Criteria: Uploaded to Inter-university Consortium for Political and Social Research (ICPSR)
URL: https://www.icpsr.umich.edu/icpsrweb/

REFERENCES:
- [Background] Hulens M, Vansant G, Claessens AL, Lysens R, Muls E. Predictors of 6-minute walk test results in lean, obese and morbidly obese women. Scand J Med Sci Sports. 2003 Apr;13(2):98-105. doi: 10.1034/j.1600-0838.2003.10273.x. PMID 12641641
- [Background] Ekkekakis P, Lind E. Exercise does not feel the same when you are overweight: the impact of self-selected and imposed intensity on affect and exertion. Int J Obes (Lond). 2006 Apr;30(4):652-60. doi: 10.1038/sj.ijo.0803052. PMID 16130028
- [Background] Williams DM. Exercise, affect, and adherence: an integrated model and a case for self-paced exercise. J Sport Exerc Psychol. 2008 Oct;30(5):471-96. doi: 10.1123/jsep.30.5.471. PMID 18971508
- [Background] Bercier KL. Effect of Weight Loss Training Protocol Using Two Different Treadmills for Obese Individuals. Boise State University Theses and Dissertations: Boise State UniversityFollow; 2014.